CLINICAL TRIAL: NCT01708135
Title: Feasibility and Efficacy of Engagement Modules for Pre-Bariatric Surgery Patients.
Brief Title: Feasibility of Use of BariCare App in Pre-bariatric Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Manpreet S. Mundi, Assistant Professor, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 12-005535
Record Dates: First submitted 2012-10-08; First posted 2012-10-16 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Smartphone Arm (Other): This is a feasibility trial and thus all participants in the study will be provided a smartphone app to assist them in preparing for bariatric surgery.
  Interventions: Behavioral: Use of smartphone app

INTERVENTIONS:
Behavioral: Use of smartphone app

SUMMARY:
This current study aims to evaluate the efficacy of engagement modules in preparing patients for bariatric surgery. With the help of the Center for Innovation (CFI), a smartphone app (Android and Apple compatible) has been created that will assist in both educating and engaging patients to develop and maintain healthy lifestyle modifications. Our goal is to create a cost-effective, smartphone-based platform that serves to not only efficiently educate but to also verify competence and keep our patients engaged during the lengthy pre-bariatric surgery process.

ELIGIBILITY:
Inclusion Criteria:

1. Patients, who upon completion of an evaluation by Endocrinology, are considered appropriate to pursue a primary, laparoscopic bariatric surgery.
2. Patients who are 18 years of age or greater.
3. Patients who own a smartphone.

Exclusion Criteria:

1. Patients with a history of a prior bariatric surgery.
2. Patients with active psychiatric disorder(s).
3. Patients with active tobacco use.
4. Patients with active substance use (alcohol, illicit drugs, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Smart phone app feasibility | 3 months
  All subjects will complete a Bariatric Surgery Questionnaire consisting of 30 questions that assess their knowldege in areas of nutrition, physical activity, and bariatric surgery. They will also be given a questionnaire on physical activity (International physical activity questionnaire or IPAQ). The primary objective is to assess improvement on both of these questionnaires with use of app.

SECONDARY OUTCOMES:
Ease of use of app | 3 months
  Through a questionnaire provided at the end of study, we will be gathering input from participants regarding ease of use of app, things they would like added or removed, as well as if they found modules helpful.

CONTACTS AND LOCATIONS:
Overall Officials: Manpreet Mundi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States